CLINICAL TRIAL: NCT07033000
Title: A Randomized, Placebo Controlled Clinical Study to Assess the Effect of a Blend of Digestive Enzymes andDandelion, Ginger & Fennel Extracts on Bloating in Adults.
Brief Title: A Randomized, Placebo Controlled Clinical Study to Assess the Effect of a Blend of Digestive Enzymes and Extracts on Bloating in Adults.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Olly, PBC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: ULOLLYBTB2
Record Dates: First submitted 2025-06-13; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Healthy
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Oral dietary supplement. Instructions: Take 1 capsule with water as needed, up to 3 capsules per day. Do not take more than 3.
  Interventions: Dietary Supplement: Placebo
- Dietary Supplement with actives (Active Comparator): Oral dietary supplement. Instructions: Take 1 capsule with water as needed, up to 3 capsules per day. Do not take more than 3.
  Interventions: Dietary Supplement: Dietary Supplement with actives

INTERVENTIONS:
Dietary Supplement: Placebo — Placebo
  Arms: Placebo
Dietary Supplement: Dietary Supplement with actives — Dietary Supplement containing blend of Digestive Enzymes, Dandelion, Ginger & Fennel Extracts
  Arms: Dietary Supplement with actives

SUMMARY:
Randomized, Double-Blind, Placebo-Controlled, Single-Center Clinical Study, where participants will take the Daily Supplement, and record Daily Symptoms, two clinical visits where Hydrogen and Methane Breath Test (HMBT) will be conducted, Abdominal Circumference Measurement will be taken, and two Self Reported Validated Questionnaires: Visual Analogue Scale (VAS) and the Quality of Life Questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Adults aged 18-65 years
2. Reported bloating and/or distention occurring at least once per week for the past 6 months, with symptoms actively present during the past 3 months
3. Willingness to avoid probiotics, antibiotics, or other supplements during the study period (unless approved by investigators)
4. Ability to provide informed consent and comply with all protocol requirements

Exclusion Criteria:

1. Diagnosed gastrointestinal diseases (e.g., inflammatory bowel disease, celiac disease, GI malignancies)
2. Use of antibiotics, laxatives, or probiotics within the past 4 weeks
3. Uncontrolled diabetes mellitus
4. Presence of mood disorders or psychiatric illness that may affect symptom perception or study compliance
5. Immunodeficiency, autoimmune conditions, or chronic inflammatory conditions
6. Excessive alcohol intake (>14 drinks/week for men, >7 drinks/week for women)
7. Use of medications known to affect gut motility or gas production (e.g., opioids, anticholinergics)
8. Pregnant or breastfeeding women
9. Use of systemic corticosteroids or immunosuppressant drugs.
10. History of reaction to the category of product tested
11. Other diseases or medications that might directly interfere in the study or put the subject's health under risk.
12. Employee of CRO or product manufacturer

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-14 (Estimated); Primary Completion 2025-08-25 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
To determine the impact of BTB on hydrogen and methane production in healthy adults | From time of enrollement to end of study at Week4
  Participants will take the Hydrogen and Methane Breath Test (HMBT) at baseline and after the study at Week4.

SECONDARY OUTCOMES:
To estimate the changes in abdominal circumference as an indicator of distention | From time of enrollement to end of study at Week4
  Standardized tape measurement at the level of the iliac crest or on top of belly button will be used to evaluate changes in abdominal distention at baseline and after the study at Week4.
To assess the changes in validated subjective questionnaire (VAS) for bloating, abdominal pain, distension, and flatulence. | From time of enrollement to end of study at Week4
  Participants will take Visual Analogue Scale (VAS) which is a self-reported assessment of bloating and distention severity using PROMIS's GI gas and bloating questionnaire at baseline and after the study at Week4.

CONTACTS AND LOCATIONS:
Locations (1):
- MusB Research, New Port Richey, Florida, United States